CLINICAL TRIAL: NCT00151255
Title: Phase III - Study on All-Trans Retinoic Acid in Combination With Standard Induction and Consolidation Therapy in Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: All-Trans Retinoic Acid in Combination With Standard Induction and Consolidation Therapy in Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard Schlenk, PD Dr., University of Ulm
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG06-04
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: age > 60 years
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; Tretinoin; Mitoxantrone

INTERVENTIONS:
Drug: Cytarabine — 100mg/m² kont. i.v. day 1-5 (induction therapy); 1000 mg/m² 2x/die i.v. day 1-3 (first consolidation cycle)
Drug: Idarubicin — 12mg/m² i.v. day 1+3 (induction therapy); 12mg/m² i.v. Tag 1+3 (second consolidation cycle)
Drug: All-trans retinoic acid — 45mg/m² p.o. day 4-6, 15mg/m² p.o. day 7-28 (induction therapy); 15mg/m² p.o. day 4-28 (consolidation therapy)
Drug: Mitoxantrone — 10mg/m² i.v. day 2-3 (first consolidation cycle)
Drug: Etoposid — 100mg/m² i.v. Tag 1-5 (second consolidation cycle)

SUMMARY:
This is a study looking at all-trans retinoic acid in combination with standard induction and consolidation therapy in older patients with newly diagnosed acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
First Induction Therapy:

* Cytarabine 100 mg/m² cont. i.v. days 1-5
* Idarubicin 12 mg/m² i.v. days 1, 3

  * ATRA 45 mg/m² p.o. days 4-6, ATRA 15 mg/m² p.o. days 7-28

Second Induction Therapy:

* Cytarabine 100 mg/m² cont. i.v. days 1-5
* Idarubicin 12 mg/m² i.v. days 1, 3

  * ATRA 45 mg/m² p.o. days 4-6, ATRA 15 mg/m² p.o. days 7-28

First Consolidation Therapy:

* Cytarabine 1000 mg/m² bid i.v. days 1-3
* Mitoxantrone 10 mg/m² i.v. days 2, 3

  * ATRA 15 mg/m² p.o. days 4-28

Second Consolidation Therapy

* Etoposide 100 mg/m² i.v. days 1-5
* Idarubicin 12 mg/m² i.v. days 1,3

  * ATRA 15 mg/m² p.o. days 4-28

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML defined according to the World Health Organization (WHO) classification (excluding acute promyelocytic leukemia [APL])
* Aged > 60 years
* All patients have to be informed about the character of the study. Written informed consent of each patient at study entry.
* Molecular and cytogenetical analyses on initial bone marrow and peripheral blood specimen have to be performed at the central reference laboratories.

Exclusion Criteria:

* Bleeding independent of the AML
* Acute promyelocytic leukemia
* Uncontrolled infection
* Participation in a concurrent clinical study
* Insufficiency of the kidneys (creatinine > 1.5 x upper normal serum level), of the liver (bilirubin, AST or AP > 2 x upper normal serum level), severe obstruction or restrictive ventilation disorder, heart failure New York Heart Association [NYHA] III/IV
* Severe neurological or psychiatric disorder interfering with ability of giving informed consent
* No consent for the registration, storage and processing of data concerning the characteristics of the AML and the individual course
* Performance status WHO > 2

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2004-06; Primary Completion 2009-06 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
event-free survival | two years

SECONDARY OUTCOMES:
kind, incidence, severity, temporal sequence and correlation of side effects of the study drugs | during therapy
complete remission (CR) rate after induction therapy | after second induction cycle
cumulative incidence of relapse | two years
cumulative incidence of death | two years
overall survival | two years

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Schlenk, Dr., Principal Investigator — University of Ulm
Locations (29):
- Austria (4):
  - Department of Hematology/Oncology, University Hospital of Innsbruck, Innsbruck
  - Department of Internal Medicine I, Krankenhaus der Barmherzigen Schwestern, Linz
  - Medical Department III, St. Johann Hospital, Salzburg
  - Center of hematology and oncology, Hanusch Hospital, Vienna
- Germany (25):
  - Department of Internal Medicine I, Central Hospital of Augsburg, Augsburg
  - Department of General Internal Medicine, University Hospital of Bonn, Bonn
  - Medical Department I, Hospital of Bremen-Mitte, Bremen
  - Department of Hematology and Oncology, Hospital Essen-Süd, Ev. Hospital of Essen-Werden, Essen
  - Department of Internal Medicine III, City Hospital Frankfurt am Main - Höchst, Frankfurt
  - Medical Department IV, University Hospital of Giessen, Giessen
  - Department of Internal Medicine, Wilhelm-Anton Hospital gGmbH, Goch
  - Centre of Internal Medicine, University Hospital of Göttingen, Göttingen
  - Department of Oncology and Hematology, University Hospital Eppendorf, Hamburg
  - Medical Department II, General Hospital Altona, Hamburg
  - Medical Department III, Hospital of Hanau, Hanau
  - Medical Department III, Hospital of Hannover-Siloah, Hanover
  - Department of Internal Medicine I, University Hospital of Saarland, Homburg
  - Medical Department II, City Hospital Karlsruhe gGmbH, Karlsruhe
  - Medical Department II, University Hospital of Kiel, Kiel
  - Department of Internal Medicine/Hematology and Oncology, Caritas Hospital Lebach, Lebach
  - Department of Hematology/Oncology, Clinical Center of Lüdenscheid, Lüdenscheid
  - Medical Department III, Clinical Center Rechts der Isar, München
  - Department of Hematology and Oncology, Clinical Center of Oldenburg gGmbH, Oldenburg
  - Department of Hematology and Oncology/Caritas Hospital St. Theresa, Saarbrücken
  - Department of Oncology, Clinical Center of Stuttgart, Stuttgart
  - Medical Department II, Diakonie Hospital, Stuttgart
  - I. Medical Department, Hospital of Barmerzigen Brüder, Trier
  - Medical Center II - Hematology/Oncology, Clinical Center Villingen-Schwenningen, Villingen-Schwenningen
  - Medical Department I, Helios Hospital Wuppertal, Wuppertal

REFERENCES:
- [Derived] Tassara M, Dohner K, Brossart P, Held G, Gotze K, Horst HA, Ringhoffer M, Kohne CH, Kremers S, Raghavachar A, Wulf G, Kirchen H, Nachbaur D, Derigs HG, Wattad M, Koller E, Brugger W, Matzdorff A, Greil R, Heil G, Paschka P, Gaidzik VI, Gottlicher M, Dohner H, Schlenk RF. Valproic acid in combination with all-trans retinoic acid and intensive therapy for acute myeloid leukemia in older patients. Blood. 2014 Jun 26;123(26):4027-36. doi: 10.1182/blood-2013-12-546283. Epub 2014 May 5. PMID 24797300
- [Derived] Schlenk RF, Taskesen E, van Norden Y, Krauter J, Ganser A, Bullinger L, Gaidzik VI, Paschka P, Corbacioglu A, Gohring G, Kundgen A, Held G, Gotze K, Vellenga E, Kuball J, Schanz U, Passweg J, Pabst T, Maertens J, Ossenkoppele GJ, Delwel R, Dohner H, Cornelissen JJ, Dohner K, Lowenberg B. The value of allogeneic and autologous hematopoietic stem cell transplantation in prognostically favorable acute myeloid leukemia with double mutant CEBPA. Blood. 2013 Aug 29;122(9):1576-82. doi: 10.1182/blood-2013-05-503847. Epub 2013 Jul 17. PMID 23863898